CLINICAL TRIAL: NCT07197619
Title: Effect of Hernia Sac Excision on Crural Tension in Paraesophageal Hernia Repair
Status: Recruiting | Type: Observational
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Amy Banks-Venegoni, Principle Investigator, Corewell Health West
Other Study IDs: 2019-732
Record Dates: First submitted 2025-02-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Paraesophageal Hernia
Keywords: Paraesophageal; Hernia
MeSH Terms: conditions — Hernia, Hiatal; Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Paraesophageal hernia can cause significant clinical symptoms, including reflux, chest pain, nausea, regurgitation, and even life threatening conditions such as bowel obstruction, and gastric volvulus. Repair of a paraesophageal hernia is associated with significant recurrence rate, with primary repair often in excess of 50%. Hernia recurrence and revisional surgery significantly increase the likelihood of complications and decreased quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18-80 undergoing elective or emergent paraesophageal hernia repair for symptomatic paraesophageal hernia will be eligible for enrollment into the study.

Exclusion Criteria:

* Patients with previous history of esophageal, gastric, diaphragmatic, or anti-reflux surgery will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Corewell Health General Surgery Patients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | Immediately following procedure
  Intraoperative Pre and Post hernia sac excision crural tension measurement will be collected.

SECONDARY OUTCOMES:
Competeness of hernia sac excision | Immediately following procedure
  Determining whether the hernia sac excision was complteted or partial
Paraesophageal hernia type | Immediately following procedure
  Comparing the paraesophageal hernia type
Mesh useage | Immediately following procedure
  Comparing the type of mesh used during the procedure
Complications | 30-days post-op
  Following patients for post-op complications
Comparing dephographics | 30-days post-op
  Looking at the patients demographics and comparing them to the above outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Corewell Health, Grand Rapids, Michigan, United States